CLINICAL TRIAL: NCT06615336
Title: Intensive Sleep Retraining and Total Sleep Deprivation for Treating Chronic Insomnia: a Randomized Controlled Trial
Brief Title: Intensive Sleep Retraining and Total Sleep Deprivation for Treating Chronic Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Charles M. Morin, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-2015
Record Dates: First submitted 2024-09-20; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Intensive Sleep Retraining; Total Sleep Deprivation; Control Condition
Keywords: chronic insomnia; intensive sleep retraining; total sleep deprivation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intensive Sleep retraining (Experimental)
  Interventions: Behavioral: Intensive Sleep retraining
- Total Sleep deprivation (Experimental)
  Interventions: Behavioral: Total Sleep Deprivation
- Control (No Intervention): The control condition consisted of one night of habitual sleep in the laboratory

INTERVENTIONS:
Behavioral: Intensive Sleep retraining — Intensive Sleep Retraining treatment consisted of 42 sleep onset trials over a 21-hour sleep deprivation period
  Arms: Intensive Sleep retraining
Behavioral: Total Sleep Deprivation — Total Sleep Deprivation treatment consisted of an equivalent 21-hour sleep deprivation period without sleep onset trials
  Arms: Total Sleep deprivation

SUMMARY:
The present study was designed to evaluate the efficacy of intensive sleep retraining for treating insomnia and explore its potential mechanisms of action. Specifically, it sought to determine whether the resolution of conditioned insomnia is the main therapeutic ingredient of intensive sleep retraining, or whether the increase in homeostatic sleep drive due to sleep deprivation accounts for sleep improvements. To isolate those two components, this study compared the short and long-term efficacy of intensive sleep retraining and total sleep deprivation for the treatment of chronic insomnia in comparison to a control condition.

DETAILED DESCRIPTION:
The pre-treatment period consisted of two consecutive weeks and was scheduled from Thursday to Thursday to coordinate the treatment period over the weekends. At the end of the pre-treatment period, participants were informed of their assignment to one of the three conditions. Participants were required to report to the sleep laboratory on Thursday at 7:00 p.m. for the night. Their time in bed was restricted to 6.5 hours (11:00 p.m. to 5:30 a.m.) to increase homeostatic sleep pressure before treatment. After waking up, participants were asked to leave the laboratory and could attend their normal daytime activities, but daytime naps were not allowed. All participants were asked to report to the laboratory at 7:00 p.m. on Friday.

Treatments

The 21-hour treatment period was scheduled from 11:00 p.m. on Friday to 8:00 p.m. on Saturday. Subjects in both the intensive sleep retraining and total sleep deprivation groups experienced at least 38.5 hours of sleep deprivation: Friday 5:30 a.m. through Saturday 8:00 p.m. Time was set aside to re-explain the protocol, answer questions, assess suicide risk again and calibrate the polysomnography montage. Participants were continuously monitored throughout the laboratory period to ensure that they were following the instructions specific to their condition. They were provided with breakfast, lunch, dinner, and snacks, but were not allowed to consume caffeine or alcohol, or to exercise. After the intensive sleep retraining and total sleep deprivation interventions, participants were not allowed to drive home for safety reasons and were instead picked up by a friend or family member or provided with a taxi voucher. There was no information about cognitive behavioral therapy for insomnia, sleep education, or sleep hygiene that was provided to any of the participants during the study.

Intensive Sleep Retraining : This treatment involved a series of 42 half-hour sleep onset opportunities repeated every 30 minutes starting at 11:00 p.m. At the beginning of each 30-minute period, participants were instructed to lie down in bed, close their eyes and relax. They were left alone in the bedroom, the lights were turned off, and the door was closed. The sleep period began when the lights were turned off. Once sleep onset was detected by the recording technician, participants were allowed to sleep for 2 to 4 consecutive minutes before being awakened. If participants did not fall asleep, the trial ended after 25 minutes, with a five-minute interval before the next sleep attempt. Participants were not given feedback about whether they fell asleep or not. Between trials, participants were instructed to get out of bed, leave the room, and either sit in a chair or stand in another room. They could talk with the experimenter or read but could not watch television or use a computer.

Total Sleep Deprivation : Participants were instructed to remain awake during the 21-hour treatment period. They could engage in quiet activities in the laboratory (e.g., reading, watching TV, using the computer) or talk with the experimenter. They could not sleep or stay in their bedrooms. A research assistant was always present to ensure that the participant did not sleep.

Control: Participants were allowed to sleep for up to 8 hours starting at 11:00 p.m. While awake, they could engage in quiet activities in the laboratory (e.g., reading, watching TV, using the computer) but were not allowed to sleep or stay in the bedroom during the day. They could attend a 1.5-hour information session about cognitive behavioral therapy for insomnia after completing the 1-month follow-up assessment.

Post-Treatment and Follow-up

Post-treatment period involved two consecutive weeks immediately after the treatment protocol. After the laboratory period, all participants were instructed to resume their normal sleep-wake schedule.

Follow-up consisted of one consecutive week of monitoring beginning 3, 7, and 11 weeks after the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years old;
* Diagnosis of chronic insomnia based on The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition criteria;
* Sleep onset latency ≥ 30 minutes for ≥ 3 nights per week for 2 weeks as measured by a daily sleep diary;
* Sleep efficiency ≤ 85% for 2 weeks as measured by a sleep diary;
* Significant distress or impairment of daytime functioning (score of at least 2 on item 5 or 7 of the Insomnia Severity Index);
* Have access to a computer with an Internet connection to complete questionnaires.

Exclusion Criteria:

* Active or unstable progressive medical condition (e.g., cancer) or degenerative neurological disease (e.g., dementia);
* Current diagnosis of major depression, dysthymia or anxiety disorders;
* Lifetime diagnosis of any psychotic or bipolar disorder;
* Other sleep disorders, sleep apnea (apnea/hypopnea index greater than 15) restless legs, or periodic limb movements during sleep (movement index with arousal greater than 15 per hour);
* Alcohol or substance use disorder in the past 12 months;
* Use of any drug known to affect sleep (e.g., cocaine) in the past 2 weeks;
* Current or planned pregnancy during the study;
* Night shift work or irregular sleep pattern (e.g., usual bedtime after 2:00 a.m. or usual wake time after 10:00 a.m.);
* Current suicidal risk;
* Body mass index greater than 32;
* Use of sleep-inducing drugs (prescription or non-prescription);
* Use of tobacco products.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | At the end of the 2-week pre-treatment; at the end of the 2-week post-treatment; and at the end of each 1-week follow-up at the 1-, 2-, and 3-month.
  7-item patient-reported measure that assessed perceived severity of sleep difficulties, daytime impairments, and distress about sleep disturbances in the past month. A higher score (0-28) indicates more severe insomnia, within four severity categories: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); severe insomnia (22-28).

SECONDARY OUTCOMES:
Visual analogue scales | During the treatment period, every hour from 8:00 a.m. to 8:00 p.m., for a total of 13 times.
  Participants were asked to circle a number from 0 to 10 corresponding to their current state on each of the following dimensions: fully awake (0) to very sleepy (10); not at all irritable (0) to very irritable (10); not at all sad (0) to very sad (10); not at all happy (0) to very happy (10); not at all angry (0) to very angry (10).
Flinders Fatigue Scale | At the end of the 2-week pre-treatment; at the end of the 2-week post-treatment; and at the end of each 1-week follow-up at the 1-, 2-, and 3-month.
  Self-reported and validated 7-item questionnaire that measured various characteristics of daytime fatigue experienced over the past two weeks. Higher scores (0-31) indicate greater fatigue.
Patient Health Questionnaire | At the end of the 2-week pre-treatment; at the end of the 2-week post-treatment; and at the end of each 1-week follow-up at the 1-, 2-, and 3-month.
  Self-reported and validated 9-item questionnaire that assessed nine symptoms of depression over the past two weeks. Total scores range from 0-27, with higher scores indicating more severe depressive symptoms, within five severity categories: none-minimal (0-4); mild (5-9); moderate (10-14); moderately severe (15-19); severe (20-27).
Generalized Anxiety Disorder Scale | At the end of the 2-week pre-treatment; at the end of the 2-week post-treatment; and at the end of each 1-week follow-up at the 1-, 2-, and 3-month.
  Self-reported and validated 7-item questionnaire that assessed seven symptoms of anxiety over the past two weeks. Total scores range from 0-21, with a higher score indicating more severe anxiety symptoms within four severity categories: minimal (0-4); mild (5-9); moderate (10-14); severe (15-21).
Actigraphy | During the 2-week pre-treatment, the 2-week post-treatment, and the 1-, 2-, and 3-month follow-ups.
  Ambulatory monitoring device that is placed on the wrist of participants to continuously record sleep-awake activity.
Sleep diary | Daily during the 2-week pre-treatment, the 2-week post-treatment, and the 1-, 2-, and 3-month follow-ups.
  Self-reported measure of the following variables: bedtime, sleep onset latency, number and duration of nighttime awakenings, wake after sleep onset, sleep quality, daytime naps, use of medication and alcohol for sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'étude des troubles du sommeil, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No